CLINICAL TRIAL: NCT03759106
Title: Optimizing a Home-based Virtual Reality Exercise Program for Chronic Stroke Patients: A Telerehabilitation Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dahlia Kairy, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIR-1319-0218
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Stroke
Keywords: Virtual reality; telerehabilitation; Stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Usual care (Other): All study participants in the control group will receive an 8-week written home exercise program (e.g. GRASP) , i.e. the usual care discharge home program.
  Interventions: Other: home written exercise program
- Experimental: Telerehabilitation system (Experimental): Participants in the experimental group will receive 8 weeks home exercise program using a virtual reality (VR) and telerehabilitation system. The intensity and choice of game for the home program will be determined by the therapist based on the patient's abilities, interests, motivation and fatigue. The patient's performance for the VR home program will be monitored asynchronously and synchronously and the program adapted to ensure it remains at an appropriate level for the patient.
  Interventions: Other: telerehabilitation/exergame system

INTERVENTIONS:
Other: home written exercise program — exercises such as picking up objects, placing objects, frequently prescribed at discharge
  Arms: No Intervention: Usual care
Other: telerehabilitation/exergame system — Video games using the Kinect camera that are carried out using the impaired arm and monitored by a therapist by videoconferencing
  Arms: Experimental: Telerehabilitation system

SUMMARY:
Stroke is a leading cause of death and long-term disability worldwide and its incidence is on the rise. Importantly, loss of arm function occurs in up to 85% of stroke survivors, with a significant long-term impact on activities of daily living, leisure activities and work. The capacity for recovery following a stroke depends on several factors, including the extent of the initial neurological damage, spontaneous recovery and rehabilitation, with possible recovery even years after the stroke. Unfortunately, accessibility of much needed rehabilitation services poststroke often remains limited, both in terms of intensity and duration, as reported in a recent report on post-stroke rehabilitation services in Quebec. Recent evidence suggests that homebased telerehabilitation (TR) is a viable approach for upper limb training post-stroke when rehabilitation services are not available. Similarly, the Canadian Best Practice Recommendations for Stroke Care update for 2013 recommends home-based patient monitoring be used when frequent monitoring is needed and face-to-face visits are not available. Hence, the investigators have developed and propose to examine the use of the VirTele system for people who have suffered a stroke who are no longer receiving rehabilitation services The VirTele system allows upper limb rehabilitation using exergames with ongoing off-line monitoring combined with online monitoring and coaching based on the self-determination theory.

DETAILED DESCRIPTION:
More specifically, the primary objective of the RCT is to provide preliminary evidence regarding efficacy of the VirTele program for upper limb motor control recovery in chronic stroke. Secondary objectives are to: i. Determine the effect of the VirTele program on upper limb function, quality of life and motivation; ii. Determine the feasibility of using the VirTele program with users at home (e.g. adherence, safety, technical difficulties, facilitators and barriers); iii. Explore the role that shared decision-making and empowerment play in exercise program adherence and progression, and in behavior modification for upper-limb use.

This study will also provide evidence of feasibility for conducting a larger-scale RCT comparing different technologies and interventions for chronic stroke rehabilitation.

A single-blind (evaluator) two-arm randomized clinical trial (RCT) is proposed for this study with participants who have had a stroke randomly allocated to: (1) 8-week training with the VirTele system.i.e. treatment group or (2) 8-week written home exercise program provided by a clinician (GRASP), i.e. exercise control group.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke (does not have to be a first time stroke);
* Mild to moderate upper limb impairment (score 2-6 Chedoke-McMaster arm component or ability to perform VR tasks at least at the lowest setting according to clinician);
* No longer receiving rehabilitation services;
* living in an area where high speed Internet access is available.

Exclusion Criteria:

* Being medically unstable;
* Severe cognitive or communication deficits;
* Visual impairments;
* Severe balance deficits limiting sitting safely independently;
* Shoulder pain limiting movements for the game;
* Previous upper limb impairment limiting potential recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Upper limb motor control at 8 weeks as measured using the Fugl-Meyer Assessment-UE (FMA-UE) | baseline and eight weeks after intervention, as well as 1 and 2 month follow up
  Upper limb motor control is assessed using a valid and reliable outcome, scores between 0-66, higher scores indicating better motor control. measure consisting of tasks to be performed by the participant

SECONDARY OUTCOMES:
Change from Baseline in Upper limb function at 8 weeks Impact on upper extremity use in daily activities will be using the Motor Activity Log, a self-reported measure of upper limb use | baseline and eight weeks after intervention, as well as 1 and 2 month follow up
  The Motor Activity Log is a questionnaire that the participant completes reporting how much the impaired upper limb is used for various daily tasks, each task is scored from 0-5 (ordinal scale, 0=do not use arm - 6=use as much as before), total score is mean of the scores.
Change from Baseline in Upper limb function at 8 weeks using the Wolf Motor Function Test | baseline and eight weeks after intervention, as well as 1 and 2 month follow up
  The Wolf Motor Function test consists of tasks that are performed by the participant with the impaired upper extremity, the tasks are rated for the quality of movement and the time taken. Items are scored on a 6 point scale, from does not attempt to movement is normal. Times tests are truncated at 120 seconds. A mean score out of a maximum of 5 is calculated.
number of sessions (feasibility) | 8 weeks (ongoing)
  number of sessions played (count)
duration of sessions (Feasibility) | 8 weeks (ongoing)
  average duration of sessions played (minutes)
Amount of time spent on the actual exe games (moving the arm) | 8 weeks (ongoing)
  amount of actual time spent using the impaired arm during the sessions (minutes)
Frequency of on-line consultations with therapist | 8 weeks (ongoing)
  Number of times real-time sessions are held between the therapist and the participant (online)
duration (minutes) of on-line consultations with therapist | 8 weeks (ongoing)
  average time spent by the therapist assisting for real-time sessions
adverse event (counts) | 8 weeks (ongoing)
  occurrence of adverse events (falls, motion sickness, dizziness, headaches) will be documented using a computerized patient log after each session.
falls (count) | 8 weeks (ongoing)
  occurrence of falls documented by the participant
adverse event - exertion (Borg Exertion Scale scored from 6-20, no exertion to maximal exertion) | 8 weeks (ongoing)
  self perceived exertion rated by the participant after the session (i.e. playing the exergame) on a scale 6-20, (no exertion to maximal exertion)

CONTACTS AND LOCATIONS:
Overall Officials: Dahlia Kairy, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Allegue DR, Kairy D, Higgins J, Archambault P, Michaud F, Miller W, Sweet SN, Tousignant M. Optimization of Upper Extremity Rehabilitation by Combining Telerehabilitation With an Exergame in People With Chronic Stroke: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2020 May 21;9(5):e14629. doi: 10.2196/14629. PMID 32097119